CLINICAL TRIAL: NCT04121520
Title: Perioperative Care of Hepatic Venous Pressure Gradient (HVPG) Measurement (CHESS1904): An International Multicenter Survey
Brief Title: Perioperative Care of HVPG Measurement (CHESS1904): An International Multicenter Survey
Status: Completed | Type: Observational
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Collaborators: LanZhou University (Other); Shandong Provincial Hospital (Other Government); Xingtai People's Hospital (Other); Zhejiang University (Other); Ankara University (Other); Chiba University Graduate School of Medicine (Unknown); Universitas Indonesia, Cipto Mangunkusumo National General Hospital (Unknown); S. Orsola-Malpighi Hospital, University of Bologna (Unknown); Universidade Federal de Pernambuco (Other); Hanyang University College of Medicine (Unknown)
Responsible Party: Principal Investigator, Xiaolong Qi, Director, Institute of Portal Hypertension, Hepatopancreatobiliary Surgery Institute of Gansu Province
Other Study IDs: CHESS1904
Record Dates: First submitted 2019-10-06; First posted 2019-10-10 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Portal Hypertension; Cirrhosis, Liver
MeSH Terms: conditions — Hypertension, Portal; Liver Cirrhosis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: At time of consent and within the same day of HVPG measurement, participants will be asked to complete a pre-operative assessment. Relevant statistics will be recorded during the HVPG procedure. Post-operative complication will also be collected and the satisfaction survey will be conducted.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — 1. Comprehensive perioperative assessment
  2. Questionnaire administration

SUMMARY:
Hepatic venous pressure gradient (HVPG) is an invasive test and requires technical skills of the operator and specialized instruments. HVPG measurement and anesthesia can cause stress responses in the body, which in turn lead to inflammatory response and immune function suppression. Thus, the perioperative care for patients undergoing HVPG measurement is crucial. This research trial studies comprehensive patient and medical worker questionnaires in predicting complications in patients with cirrhosis undergoing HVPG measurement. Comprehensive patient and medical worker questionnaires may help identify complications, such as the need for assistance in taking medication, decreased mobility and released tension that may improve outcomes.

DETAILED DESCRIPTION:
Portal hypertension is an important factor affecting the clinical outcomes of cirrhosis patients, and its severity determines the occurrence of development of cirrhosis complications, such as rupture and bleeding of gastroesophageal varices, ascites, and hepatorenal syndrome. The direct measurement of portal pressure is an extremely invasive and high-risk procedure. In addition, changes in intra-abdominal pressure will affect the portal pressure, which leads to unreliable results. The hepatic venous pressure gradient (HVPG) is the difference between wedged hepatic venous pressure and free hepatic venous pressure and reflects the pressure difference between the hepatic portal vein and the intra-abdominal veins. In recent years, the status of HVPG in clinical application of cirrhotic portal hypertension has gradually improved. In 2016, the American Association for the Study of Liver Diseases (AASLD) issued a consensus on risk stratification, diagnosis, and management of portal hypertensive bleeding in cirrhosis and re-emphasized the value of HVPG in assessing the cirrhosis staging, occurrence of complications and treatment goals. However, HVPG is an invasive test and requires technical skills of the operator and specialized instruments. HVPG measurement and anesthesia can cause stress responses in the body, which in turn lead to inflammatory response and immune function suppression. Thus, the perioperative care for patients undergoing HVPG measurement is crucial. This research trial studies comprehensive patient and medical worker questionnaires in predicting complications in patients with cirrhosis undergoing HVPG measurement. Comprehensive patient and medical worker questionnaires may help identify complications, such as the need for assistance in taking medication, decreased mobility and released tension that may improve outcomes.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants must meet the following criteria:

1. aged between 18-75 years, no restriction on gender;
2. clinically and/or pathologically diagnosed sinusoidal cirrhosis;
3. with written informed consent
4. scheduled to undergo HVPG measurement according to the following indications: 1) assessment of the efficacy of primary and secondary prophylactic drugs for gastroesophageal variceal bleeding; 2) predicting the risk of gastroesophageal variceal bleeding and guiding the selection of the treatment regimens; 3) predicting of risk, progression, and clinical outcomes of decompensation events in cirrhosis; 4) evaluation of the efficacy of new drugs; 5) evaluation of the accuracy of new non-invasive techniques; diagnosis and differential diagnosis of types of portal hypertension.

Exclusion Criteria:

Those cases that meet any of the following criteria should be excluded:

1. contradictions for HVPG measurement;
2. pregnant or lactating woman;
3. severe coagulopathy (international normalized ratio>5);
4. severe heart, lung, or kidney disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with cirrhosis who were scheduled to undergo HVPG measurement
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Post-operative satisfaction | 1 day
  After the procedure of HVPG (within the same day), participants will be asked to complete a pain scale which was experienced during and after the HVPG procedure. The pain scale ranges from 0 to 10 with 0 representing 'not at all' and 10 representing 'excessively'.

SECONDARY OUTCOMES:
Pre-operative perception | 1 day
  At time of consent and within the same day of HVPG procedure, participants will be asked to complete a pain scale which was felt to be experienced during the HVPG procedure. The pain scale ranges from 0 to 10 with 0 representing 'not at all' and 10 representing 'excessively'.
Number of intra-operative complications | 1 day
  Number of complications (e.g. vasovagal reflex, arrhymia, inadvertent arterial puncture, hypersensitivity to contrast agents, pneumothorax) happened during the HVPG procedure.
Number of post-operative complications | 1 day
  Number of complications (e.g. bleeding at the puncture point, contrast-induced nephropathy, infection, jugular vein thrombosis) happened after the HVPG procedure.
Methods selection of HVPG measurement | 1 day
  Including the selection of routes for insertion of catheter, hepatic vein used for the assessment and the angiographic catheter used during the HVPG procedure.
The result of HVPG measurement | 1 day
  The mean value of HVPG measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolong Qi, M.D., Principal Investigator — LanZhou University; Necati Örmeci, M.D., Principal Investigator — Ankara University
Locations (10):
- Universidade Federal de Pernambuco, Recife, Brazil
- China (4):
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Xingtai People's Hospital, Xingtai, Hebei
  - Shandong Provincial Hospital affiliated to Shandong University, Jinan, Shandong
  - The First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
- Universitas Indonesia, Cipto Mangunkusumo National General Hospital, Jakarta, Indonesia
- S. Orsola-Malpighi Hospital, University of Bologna, Bologna, Italy
- Chiba University Graduate School of Medicine, Chiba, Japan
- Hanyang University College of Medicine, Seoul, South Korea
- Ankara University School of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] de Franchis R; Baveno VI Faculty. Expanding consensus in portal hypertension: Report of the Baveno VI Consensus Workshop: Stratifying risk and individualizing care for portal hypertension. J Hepatol. 2015 Sep;63(3):743-52. doi: 10.1016/j.jhep.2015.05.022. Epub 2015 Jun 3. No abstract available. PMID 26047908
- [Background] Garcia-Tsao G, Abraldes JG, Berzigotti A, Bosch J. Portal hypertensive bleeding in cirrhosis: Risk stratification, diagnosis, and management: 2016 practice guidance by the American Association for the study of liver diseases. Hepatology. 2017 Jan;65(1):310-335. doi: 10.1002/hep.28906. Epub 2016 Dec 1. No abstract available. PMID 27786365
- [Background] Bosch J, Abraldes JG, Berzigotti A, Garcia-Pagan JC. The clinical use of HVPG measurements in chronic liver disease. Nat Rev Gastroenterol Hepatol. 2009 Oct;6(10):573-82. doi: 10.1038/nrgastro.2009.149. Epub 2009 Sep 1. PMID 19724251
- [Background] Qi X, Berzigotti A, Cardenas A, Sarin SK. Emerging non-invasive approaches for diagnosis and monitoring of portal hypertension. Lancet Gastroenterol Hepatol. 2018 Oct;3(10):708-719. doi: 10.1016/S2468-1253(18)30232-2. PMID 30215362